CLINICAL TRIAL: NCT01264367
Title: A Study to Evaluate the Efficacy and Safety of Clevudine and Peg-interferon in Sequence Compared With Clevudine Alone in the Patients With HBeAg(+) Chronic Hepatitis B or Clevudine and Peg-interferon Sequential Treatment in Patients With Chronic Hepatitis B Who Have HBeAg(+)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bukwang Pharmaceutical (Industry)
Responsible Party: Bukwang Pharm.CO.,LTD, Bukwang Pharm.CO.,LTD
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CMC-403; CMC-403
Record Dates: First submitted 2010-12-19; First posted 2010-12-21 (Estimated); Last update posted 2014-12-18 (Estimated); Status verified 2012-07

CONDITIONS: HBeAg(+) Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — clevudine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Clevudine 30mg
  Interventions: Drug: Clevudine
- 2 (Active Comparator): Clevudine 30mg + peg-interferon 180mcg
  Interventions: Drug: Clevudine + Peg-interferon

INTERVENTIONS:
Drug: Clevudine — 30mg,QD
  Other Names: Levovir
  Arms: 1
Drug: Clevudine + Peg-interferon — 30mg, QD(for 24 weeks) + 180mcg,QW(for 24 weeks)
  Other Names: Levovir + Pagasys
  Arms: 2

SUMMARY:
A study to evaluate the efficacy and safety of clevudine and peg-interferon in sequence compared with clevudine alone in the patients with HBeAg(+) chronic Hepatitis B or clevudine and peg-interferon sequential treatment in patients with chronic Hepatitis B who have HBeAg(+)

ELIGIBILITY:
Inclusion Criteria:

1. Patient is between 18~60 years
2. Patient is HBV DNA positive with DNA levels ≥ 5 x 10^5 copies/mL within 30 days of baseline.
3. Patient is documented to be HBsAg positive for > 6 months and Patient is HBeAg positive.
4. Patient has ALT levels >=80IU/L, prothrombin time(INR)<1.7 and a serum albumin level of at least 3.5 g/dL.
5. Patient has hemoglobin levels >=11.5g/dl(if woman) or >=12.5g/dl(if man)
6. Women of childbearing potential must have a negative urine pregnancy test(β-HCG) taken within 14 days of starting therapy.
7. Patient is able to give written informed consent prior to study start and to comply with the study requirements.

Exclusion Criteria:

1. Patient is currently receiving antiviral, immunomodulatory, cytotoxic or corticosteroid therapy.
2. Patients previously treated with interferon, peg-interferon, clevudine, lamivudine, adefovir, entecavir, telbivudine, tenofovir or any other investigational nucleoside for HBV infection.
3. Patient is coinfected with HCV or HIV.
4. Patient with clinical evidence of decompensated liver disease or HCC
5. Patient has WBC levels < 3.0x10^9/L
6. Patient has Platelets levels < 90x10^9/L
7. Patient has alpha fetoprotein levels > 100ng/mL
8. Patient has a history of Thyroid disease.
9. Patient has a history of autoimmune hepatitis.
10. Patient is pregnant or breast-feeding.
11. Patient is unwilling to use an "effective" method of contraception during the study and for up to 3 months after the use of study drug ceases.
12. Patient has a clinically relevant history of abuse of alcohol or drugs.
13. Patient has a significant immunocompromised, gastrointestinal, renal, hematological, psychiatric, bronchopulmonary, biliary diseases excluding asymptomatic GB stone, neurological, cardiac, oncologic or allergic disease or medical illness that in the investigator's opinion might interfere with therapy. The patient with a benign tumor, excluded if judged by an investigator that the continuation of study would be interfered by the tumor.
14. Patient has creatinine clearance less than 60mL/min as estimated by the following formula: (140-age in years) (body weight [kg])/(72) (serum creatinine [mg/dL]) [Note: multiply estimates by 0.85 for women]

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2008-12; Primary Completion 2013-08 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
antiviral activity;Proportion of patients with HBV DNA below LOD(HBV DAN levels < 300 copies/mL) by real time PCR | At week 48

SECONDARY OUTCOMES:
antiviral activity;Proportion of patients with HBV DNA below LOD(HBV DAN levels < 300 copies/mL) by real time PCR | At week 72
antiviral activity: The change of HBV DNA from the baseline | Screening, Day1(predose), at week 12, 24, 36, 48, 60, 72
ALT normalization rate | Screening, Day1(predose), at week 12, 24, 36, 48, 60, 72
Proportion sustained complete response of patients with complete response | At week 72
Immunological endpoints | Day1(predose), at week 24, 48, 72
Proportion of patients with HBeAg loss/ HBeAg seroconversion | At week 48

CONTACTS AND LOCATIONS:
Overall Officials: Lee Chang Don, MD, PhD, Principal Investigator — The catholic university of korea, Uijeongbu ST.Mary's hospital
Locations (1):
- Uijeongbu St.Mary's Hospital, Uijeongbu-si, South Korea